CLINICAL TRIAL: NCT05219110
Title: Hyperhydration to Improve Kidney Outcomes in Children With Shiga Toxin-Producing E. Coli Infection: A Multinational Embedded Cluster Crossover Randomized Trial
Brief Title: Hyperhydration in Children With Shiga Toxin-Producing E. Coli Infection
Acronym: HIKO-STEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Children's Hospital Medical Center, Cincinnati (Other); Washington University School of Medicine (Other); University of Utah (Other); Seattle Children's Hospital (Other); University of Colorado, Denver (Other); Emory University (Other); University of California, Davis (Other); Baylor College of Medicine (Other); Indiana University School of Medicine (Other); University of Alabama at Birmingham (Other); Arkansas Children's Hospital Research Institute (Other); Children's National Research Institute (Other); Children's Hospitals and Clinics of Minnesota (Other); Medical University of South Carolina (Other); University of Louisville (Other); University of Oklahoma (Other); Oregon Health and Science University (Other); University of California, San Diego (Other); McMaster University (Other); The Hospital for Sick Children (Other); University of Alberta (Other); University of Kentucky (Other); Case Western Reserve University (Other); Nationwide Children's Hospital (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DMID 21-0042; R01AI165327 (NIH)
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-12

CONDITIONS: Shiga Toxin-Producing Escherichia Coli (E. Coli) Infection; Hemolytic-Uremic Syndrome
Keywords: Child; Hemolytic Uremic Syndrome; Shiga-Toxigenic Escherichia coli; Renal Replacement Therapy; Acute Kidney Injury; Ambulatory Care; Emergency Department
MeSH Terms: conditions — Escherichia coli Infections; Infections; Hemolytic-Uremic Syndrome; Acute Kidney Injury; Emergencies | interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Cluster crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperhydration (Experimental): In this study arm, all eligible children are admitted for the administration of intravenous fluids.
  The following specifics will form the basis of the fluid management protocol:
  1. Reversal of dehydration: Initial ED rehydration strategies should focus on rapidly reversing dehydration.
  2. Infusion of 200% of maintenance fluids x 24 hours
  3. If hematocrit reduction < 20% from initial value, repeat step #2 [infusion of 200% maintenance fluids x 24 hours].
  4. Oral fluids permitted ad lib.
  5. Once the target hematocrit reduction is achieved (20% decrement in initial HCT) AND a 10% weight gain, adjust total IV fluid volume to maintain targeted weight gain: insensible plus output (i.e., urine plus stool).
  Interventions: Other: Infusion of 200% maintenance fluids as balanced crystalloid IV solution
- Conservative Fluid Management (Active Comparator): The conservative fluid management arm has been designed to align and integrate into existing local practice patterns. Implementation of this approach will allow institutions and their practitioners to choose their management of protocol eligible children. All children will undergo a protocolized baseline evaluation that includes reversal of dehydration (if present) and follow-up plan (see Pre-Pathway care). The fluid management decision in the ED (i.e., to treat dehydration) will be at the discretion of the clinical care team. In the absence of evidence of microangiopathy (i.e., normal urinalysis, LDH, hemoglobin and platelet counts, and creatinine concentrations), the decision to admit the child to hospital or discharge the child to home will be at the discretion of the clinical care team. If microangiopathy is present (i.e., abnormal urinalysis, LDH, hemoglobin or platelet counts, or creatinine concentrations) admission for monitoring will be required.
  Interventions: Other: Oral fluids; infusion of up to 110% maintenance fluids as balanced crystalloid IV solution

INTERVENTIONS:
Other: Infusion of 200% maintenance fluids as balanced crystalloid IV solution — Infusion of 200% of maintenance fluids x 24 hours provided, ideally, as a balanced crystalloid (PlasmaLyteTM, Ringer's Lactate) IV solution. Electrolytes and dextrose may be administered as required and desired by the clinical care team; customized solutions are permitted if so desired. Intravenous fluid solutions containing < 130 mEq/L sodium may increase risk for hyponatremia and may be less effective in achieving intravascular volume expansion and should be avoided.
  Arms: Hyperhydration
Other: Oral fluids; infusion of up to 110% maintenance fluids as balanced crystalloid IV solution — Administration of less than or equal to 110% of maintenance fluids as oral or balanced crystalloid IV solution.
  Arms: Conservative Fluid Management

SUMMARY:
The objective of this study is to determine if early high volume intravenous fluid administration (hyperhydration) may be effective in mitigating or preventing complications of shiga toxin-producing E. coli (STEC) infection in children and adolescents when compared with traditional approaches (conservative fluid management).

DETAILED DESCRIPTION:
The hemolytic uremic syndrome (HUS) is the most serious complication of high-risk Shiga toxin-producing Escherichia coli (STEC) infection and the most common cause of acquired acute kidney injury in otherwise healthy children. HUS develops in up to 20% of children following STEC infection, 60% of whom require temporary renal replacement therapy (RRT); an additional 50% develop serious extrarenal complications. Although mortality from acute HUS is low (1-3%), it has remained constant for three decades and approximately 30% of HUS survivors experience long-term sequelae, chiefly chronic kidney disease, hypertension, and diabetes. There have been only three relatively small, randomized trials to prevent progression to HUS and/or to reduce kidney injury once HUS is established; none have demonstrated benefits, and none have been performed since 1999.

Recent cohort studies suggest that early intravascular volume expansion (hyperhydration) in STEC infected children could be nephroprotective if and when HUS occurs. However, more evidence is needed before hyperhydration supplants traditional 'wait and see' (i.e., conservative fluid management) reactive care approaches which focus on outpatient care and minimizing intravenous fluid administration to avoid fluid overload in children who do develop HUS. Here, we will confirm or refute the hypothesis that aggressive volume expansion, administered early in STEC infected children, is associated with better renal outcomes and fewer adverse events than conservative management by accomplishing three Specific Aims: (1) Determine the effectiveness of hyperhydration in decreasing the prevalence of Major Adverse Kidney Events by 30 days (defined as death, RRT, or sustained loss of kidney function at 30 days) in STEC-infected children versus conservative fluid management; (2) Determine the effectiveness and safety of hyperhydration in decreasing HUS and life-threatening, extrarenal complications in STEC-infected children versus conservative fluid management; (3) Create a biorepository that will be linked to our clinical data to identify prognostic biomarkers and therapeutic targets in STEC-infected children.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study (i.e., to be enrolled in the relevant institutional clinical care pathway), an individual must meet all of the following criteria:

1. Aged 9.0 months to <21 years at the time of informed consent.
2. Evidence of high-risk STEC infecting pathogen defined by any of the following:

   1. Bloody diarrhea within the preceding 7 days

      * Positive STEC culture OR
      * Positive antigen/polymerase chain reaction test for toxin/gene type not otherwise specified OR
   2. Bloody or Non-bloody diarrhea within the preceding 7 days

      •Presumptive diagnosis of HUS
      * (meeting all 3 HUS criteria - anemia, thrombocytopenia, and renal insufficiency) OR
   3. Non-bloody or no diarrhea

      * Positive STEC culture for high-risk strain (i.e., O103, O104, O111, O113, O121, O145 or O157) OR
      * Positive antigen/polymerase chain reaction test Stx2 toxin/gene

Exclusion Criteria:

All individuals meeting any of the exclusion criteria at baseline will be excluded from study participation.

1. Presence of Advanced HUS defined by:

   1. Hematocrit <30% AND
   2. Platelet count <150 x 103/mm3 AND
   3. Creatinine > 2.0 mg/dL (177 µmol/L)

      * The presence of only 1 or 2 of these criteria will not result in patient exclusion, regardless of how close the 3rd criterion is to meeting the exclusion criteria.
2. Prior episode of HUS or diagnosis of atypical HUS.
3. Chronic disease limiting fluid volumes administered (e.g. impaired renal, liver, or cardiac function, chronic lung disease).
4. Evidence of anuria (i.e., no urine output for > 24 hours).
5. Hypoxemia requiring oxygen therapy
6. Hypertensive emergency
7. Greater than or equal to 10 days since onset of diarrhea or if no diarrhea then the onset of other symptoms.
8. Patients with known pregnancy
9. Patients or caregivers with language barriers impairing appropriate conduct of the study protocol.

Ages: 9 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1040 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Kidney Events by 30 days (MAKE30) | 30 days
  1. Death due to any cause censored at 30 days after enrollment OR
  2. Provision of RRT, any modality, within 30 days of trial enrollment OR
  3. Sustained loss of kidney function (100% increase of serum sCr from baseline at 30±7 days)

SECONDARY OUTCOMES:
Number of Participants with Significant Extrarenal Complications (life-threatening): | 30 days
  a. Neurologic: i. Seizures requiring anticonvulsant therapy ii. Coma iii. Thrombotic or hemorrhagic stroke confirmed by neuroimaging b. Cardiac: i. Myocardial infarction ii. Myocarditis iii. Myocardial dysfunction iv. Arrhythmias requiring cardioversion or pharmacological anti-arrhythmic therapy c. Respiratory: i. Respiratory failure ii. Pleural effusions d. Gastrointestinal: i. Hyperglycemia requiring prolonged insulin therapy ii. Bowel obstruction/perforation requiring surgical repair iii. Intussusception requiring reduction iv. Acute cholecystitis v. Pancreatitis vi. Hepatitis/ liver failure vii. Ascites requiring paracentesis e. Infectious complications i. Bacteremia ii. Peritonitis
Number of Participants who Develop HUS among those without it at randomization | 30 days
  1. Anemia (hematocrit level <30%) AND
  2. Thrombocytopenia (platelet count <150 X 103/mm3) AND
  3. Renal azotemia (serum creatinine concentration >upper limit of reference range for age)

OTHER OUTCOMES:
Length of Stay | 30 days
  1. Number of days as an inpatient
  2. Number of days in an intensive care unit (a unit capable of providing mechanical ventilation)
  3. Hospital-Free Days: Measured as the number of calendar days alive and out of the hospital between randomization (day 0) and day 30. Patients who die prior to hospital discharge will be recorded as zero hospital-free days.
  4. Score each hospital day
     * # days with HUS with RRT
     * # days with HUS without RRT
     * # days in hospital - no HUS
Number of Participants who Receive Transfusion Therapy | 30 days
  1. Red Blood Cell
  2. Platelets
Number of Participants who Receive Invasive Medical Procedures | 30 days
  1. Mechanical ventilation
  2. Endotracheal intubation
  3. Thoracentesis, thoracotomy, ARDS
  4. Central venous catheter insertion
  5. Dialysis catheter insertion
  6. Therapeutic plasma exchange
  7. Other operative room surgical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MDCM, Principal Investigator — University of Calgary
Locations (26):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, San Diego, La Jolla, California
  - University of California, Davis, Sacramento, California
  - University of Colorado Denver, Denver, Colorado
  - Children's Research Institute, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Indiana University Children's Hospital, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Minnesota Hospital, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - McMaster University, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imdad A, Nelson JR, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2025 Apr 25;4(4):CD012997. doi: 10.1002/14651858.CD012997.pub3. PMID 40277027
- [Derived] Freedman SB, Schnadower D, Estes M, Casper TC, Goldstein SL, Grisaru S, Pavia AT, Wilfond BS, Metheney M, Kimball K, Tarr PI; Hyperhydration to Improve Kidney Outcomes in children with Shiga Toxin-producing E. Coli infection (HIKO-STEC) Study Team. Hyperhydration to Improve Kidney Outcomes in Children with Shiga Toxin-Producing E. coli Infection: a multinational embedded cluster crossover randomized trial (the HIKO STEC trial). Trials. 2023 May 27;24(1):359. doi: 10.1186/s13063-023-07379-w. PMID 37245030